CLINICAL TRIAL: NCT01625455
Title: Effect of Neurokinin-1 Receptor (NK1R) Antagonism on Pruritus in Patients With Sezary Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, Chair and Physician-in-chief, Department of Medicine, Hugh Jackson Morgan Professor Medicine and Pharmacology, Vanderbilt University School of Medicine, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110806
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Sezary Syndrome; Pruritus
Keywords: Sezary Syndrome; Pruritus; Aprepitant; Neurokinin-1
MeSH Terms: conditions — Sezary Syndrome; Pruritus | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant (Active Comparator): Aprepitant will be given orally in a dose of 125mg on day 1 and 80mg daily on each subsequent day for a total of 7 days.
  Interventions: Drug: Aprepitant
- Placebo (Placebo Comparator): Matching placebo will be given in place of aprepitant
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — Aprepitant will be given orally in a dose of 125mg on day 1 and 80mg daily on each subsequent day for a total of 7 days.
  Other Names: Emend
  Arms: Aprepitant
Drug: Placebo — Placebo will be given orally for a total of 7 days.
  Arms: Placebo

SUMMARY:
The purpose of this randomized, double-blinded, placebo-controlled study is to test the hypothesis that administration of aprepitant will decrease the severity of pruritus in patients with Sèzary Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Known Sezary Syndrome
* Pruritus uncontrolled by conventional treatment. Baseline visual analogue scale > 4.
* Age 18 through 80 years of age.
* Stable medication regimens for both Sezary Syndrome and pruritus for 3 months prior to study participation.

Exclusion Criteria:

* Known hepatic impairment (defined as liver function tests >3 times the upper limit of normal).
* Pregnancy (all women of child-bearing potential will undergo urine beta-hcg testing).
* Concurrent use of pimozide, terfenadine, astemizole, or cisapride.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-02; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Bernengo MG, Novelli M, Quaglino P, Lisa F, De Matteis A, Savoia P, Cappello N, Fierro MT. The relevance of the CD4+ CD26- subset in the identification of circulating Sezary cells. Br J Dermatol. 2001 Jan;144(1):125-35. doi: 10.1046/j.1365-2133.2001.04014.x. PMID 11167693
- [Background] Booken N, Heck M, Nicolay JP, Klemke CD, Goerdt S, Utikal J. Oral aprepitant in the therapy of refractory pruritus in erythrodermic cutaneous T-cell lymphoma. Br J Dermatol. 2011 Mar;164(3):665-7. doi: 10.1111/j.1365-2133.2010.10108.x. Epub 2011 Jan 28. No abstract available. PMID 21039410
- [Background] Duval A, Dubertret L. Aprepitant as an antipruritic agent? N Engl J Med. 2009 Oct 1;361(14):1415-6. doi: 10.1056/NEJMc0906670. No abstract available. PMID 19797294
- [Background] Cevikbas F, Steinhoff M, Ikoma A. Role of spinal neurotransmitter receptors in itch: new insights into therapies and drug development. CNS Neurosci Ther. 2011 Dec;17(6):742-9. doi: 10.1111/j.1755-5949.2010.00201.x. Epub 2010 Oct 15. PMID 20950328
- [Background] Lambeir AM, Durinx C, Scharpe S, De Meester I. Dipeptidyl-peptidase IV from bench to bedside: an update on structural properties, functions, and clinical aspects of the enzyme DPP IV. Crit Rev Clin Lab Sci. 2003 Jun;40(3):209-94. doi: 10.1080/713609354. PMID 12892317
- [Background] Ahmad S, Wang L, Ward PE. Dipeptidyl(amino)peptidase IV and aminopeptidase M metabolize circulating substance P in vivo. J Pharmacol Exp Ther. 1992 Mar;260(3):1257-61. PMID 1372050
- [Background] Heymann E, Mentlein R. Liver dipeptidyl aminopeptidase IV hydrolyzes substance P. FEBS Lett. 1978 Jul 15;91(2):360-4. doi: 10.1016/0014-5793(78)81210-1. No abstract available. PMID 680144
- [Background] Mussap CJ, Geraghty DP, Burcher E. Tachykinin receptors: a radioligand binding perspective. J Neurochem. 1993 Jun;60(6):1987-2009. doi: 10.1111/j.1471-4159.1993.tb03484.x. PMID 8388031
- [Background] Hesketh PJ. Chemotherapy-induced nausea and vomiting. N Engl J Med. 2008 Jun 5;358(23):2482-94. doi: 10.1056/NEJMra0706547. No abstract available. PMID 18525044
- [Background] Olsen E, Vonderheid E, Pimpinelli N, Willemze R, Kim Y, Knobler R, Zackheim H, Duvic M, Estrach T, Lamberg S, Wood G, Dummer R, Ranki A, Burg G, Heald P, Pittelkow M, Bernengo MG, Sterry W, Laroche L, Trautinger F, Whittaker S; ISCL/EORTC. Revisions to the staging and classification of mycosis fungoides and Sezary syndrome: a proposal of the International Society for Cutaneous Lymphomas (ISCL) and the cutaneous lymphoma task force of the European Organization of Research and Treatment of Cancer (EORTC). Blood. 2007 Sep 15;110(6):1713-22. doi: 10.1182/blood-2007-03-055749. Epub 2007 May 31. PMID 17540844
- [Background] Vonderheid EC, Bernengo MG, Burg G, Duvic M, Heald P, Laroche L, Olsen E, Pittelkow M, Russell-Jones R, Takigawa M, Willemze R; ISCL. Update on erythrodermic cutaneous T-cell lymphoma: report of the International Society for Cutaneous Lymphomas. J Am Acad Dermatol. 2002 Jan;46(1):95-106. doi: 10.1067/mjd.2002.118538. PMID 11756953
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956
- [Derived] Zic JA, Straka BT, McGirt LY, Nian H, Yu C, Brown NJ. Aprepitant for the Treatment of Pruritus in Sezary Syndrome: A Randomized Crossover Clinical Trial. JAMA Dermatol. 2018 Oct 1;154(10):1221-1222. doi: 10.1001/jamadermatol.2018.2510. PMID 30140912

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seven subjects were consented and enrolled. Two did not meet inclusion/exclusion criteria and were not randomized.
Groups:
- Placebo Then Aprepitant: These subjects received placebo during the first week and then crossed over to aprepitant for the second week.
- Aprepitant Then Placebo.: These subjects received aprepitant during the first week and then crossed over to placebo for the second week.
Period: Overall Study
Arm/Group | Placebo Then Aprepitant | Aprepitant Then Placebo.
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Aprepitant | Aprepitant Then Placebo. | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 71 [66 to 76] | 58.3 [47 to 77] | 63.4 [47 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Severity of Pruritus
Description: The primary endpoint is the severity of pruritus as measured on the visual analogue scale. A score of 100 indicated the worst pruritus imaginable, while 0 indicated no pruritus.
Time Frame: one week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | 58.20 (17.82) | 47.47 (20.22)

2. Secondary Outcome: Quality of Life
Description: The secondary endpoint is the quality of life as measured on the Dermatology Quality of Life Index (DLQI).
  For a series of 10 questions the responses are scored: Very much, scored 3; A lot, scored 2; A little, scored 1; Not at all, scored 0; Not relevant, scored 0; and Question unanswered, scored 0. The scores are summed and the larger the score the greater the effect of the dermatological disease impact on quality of life.
  Maximum response for all ten questions 30, minimum 0.
Time Frame: one week
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 5 | 5
scores on a scale | 14.2 (9.7) | 14.8 (10.3)

ADVERSE EVENTS:
Arm/Group | Placebo | Aprepitant
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes